CLINICAL TRIAL: NCT01118377
Title: A Phase II Trial of Capecitabine Rapidly Disintegrating Tablets and Concomitant Radiation Therapy in Children With Newly Diagnosed Brainstem Gliomas
Brief Title: A Study of Capecitabine (Xeloda®) and Concomitant Radiation Therapy in Children With Newly Diagnosed Brainstem Gliomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Pediatric Brain Tumor Consortium (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NO21125; PBTC-030
Record Dates: First submitted 2010-04-15; First posted 2010-05-06 (Estimated); Results first posted 2013-12-03 (Estimated); Last update posted 2014-02-06 (Estimated); Status verified 2014-02

CONDITIONS: Brainstem Glioma
MeSH Terms: interventions — Capecitabine; Radiotherapy

ARMS (1):
- Capecitabine + radiation therapy (Experimental): Participants received 9 weeks of capecitabine 650 mg/m^2 orally (po) twice daily (bid) plus radiation therapy (180 cGy/day 5 days a week, total target dose of 56 Gy) followed by a 2-week rest period. Participants then received 3 cycles of capecitabine 1250 mg/m^2 po bid for 14 days followed by a 7-day rest period without radiation therapy.
  Interventions: Drug: Capecitabine; Radiation: Radiation therapy

INTERVENTIONS:
Drug: Capecitabine — Capecitabine was supplied as film-coated tablets.
  Other Names: Xeloda
Radiation: Radiation therapy — Local irradiation using conformal, volume-based delivery techniques. The nominal energy of the X-rays was ≥ 4 MV.

SUMMARY:
This study evaluated the effect of capecitabine and concomitant radiation therapy in children with newly diagnosed brainstem gliomas.

DETAILED DESCRIPTION:
The open-label phase 2 study NO21125 (NCT01118377) evaluated the progression-free survival, safety, and pharmacokinetics of capecitabine (Xeloda®) rapidly disintegrating tablets and concomitant radiation therapy in children and adolescent patients with newly diagnosed brainstem glioma. There were 2 phases to the study: A 9-week radiation phase, followed by a 2-week rest period, and a 9-week post-radiation phase. In the radiation phase, capecitabine 650 mg/m^2 was administered orally twice daily for 9 weeks. Concomitantly, patients received radiation therapy (180 cGy fractions) 5 days a week for a total target dose of 56 Gy. During the 9-week post-radiation phase of the study, capecitabine 1250 mg/m^2 was administered orally twice daily for 14 days followed by a 7-day rest period. This cycle of 14 days treatment followed by 7 days rest was repeated 2 additional times. The dose could be adjusted according to toxicity and body surface area.

The single-arm phase 1 study NO18517 (NCT00532948) assessed the maximum tolerated dose and dose-limiting toxicities of capecitabine (Xeloda®) administered concurrently with radiation therapy in children with newly diagnosed diffuse intrinsic brain stem gliomas and high grade gliomas. Patients in the phase 1 study NO18517 who were diagnosed with intrinsic brainstem glioma and who were treated at the established maximum tolerated dose of capecitabine 650 mg/m^2/dose twice a day were included in the analyses of the phase 2 study NO21125.

The efficacy and safety results of study NO21125 are reported below.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric and adolescent patients ≥ 3 to < 18 years of age.
* Patients must have a newly diagnosed non-disseminated intrinsic infiltrating brainstem glioma.
* Karnofsky Performance Scale (if > 16 years of age) or Lansky Performance Score (if ≤ 16 years of age) ≥ 50% assessed within 2 weeks prior to registration to study.
* Patients must not have received any prior chemotherapy or bone marrow transplant for the treatment of brainstem glioma. Prior dexamethasone and/or surgery are allowed.
* Adequate organ function.

Exclusion Criteria:

* Patients receiving any other anticancer or experimental drug therapy.
* Patients with uncontrolled infection.
* Known dihydropyrimidine dehydrogenase (DPD) deficiency.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2007-05; Primary Completion 2013-01 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (8):
- United States (8):
  - San Francisco, California
  - Washington D.C., District of Columbia
  - Chicago, Illinois
  - Durham, North Carolina
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Memphis, Tennessee
  - Houston, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Capecitabine + Radiation Therapy
Started | 45
Completed | 3
Not Completed | 42
Not completed — Did Not Receive Study Medication | 1
Not completed — Death | 38
Not completed — Failure to Return | 3

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population: All enrolled participants who received at least 1 dose of capecitabine. One of the 45 participants did not receive treatment and was not included in the intent-to-treat population (34 participants from study NO21125 and 10 participants from study NO18517).
Arm/Group | Capecitabine + Radiation Therapy
Number analyzed (Participants) | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.5 (3.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 22

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Progression-free survival was defined as the time from the initiation of treatment to the earliest date of failure (disease progression, death from any cause, or a second malignancy) or to the last assessment date for patients who did not fail. Disease progression was defined as progressive neurologic abnormalities or worsening neurologic status not explained by causes unrelated to tumor progression (eg, anticonvulsant or corticosteroid toxicity, electrolyte disturbances, sepsis, hyperglycemia, weaning of steroids, radiation necrosis, etc); or a greater than 25% increase in the bi-dimensional measurement of the tumor, as compared with the previous scan; or the appearance of a new lesion; or an increase in the doses of dexamethasone required to maintain stable neurologic status or imaging.
Time Frame: Baseline to the end of the study (up to 20 weeks)
Population: Intent-to-treat population: All enrolled participants who received at least 1 dose of capecitabine.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Capecitabine + Radiation Therapy
Number analyzed (Participants) | 44
Months | 4.9 [4.5 to 6.0]

2. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from the initiation of therapy to the date of death from any cause or to the date the patient was last known to be alive for surviving patients.
Time Frame: Baseline to the end of the study (up to 20 weeks)
Population: Intent-to-treat population: All enrolled participants who received at least 1 dose of capecitabine.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Capecitabine + Radiation Therapy
Number analyzed (Participants) | 44
Months | 10.3 [7.7 to 12.9]

3. Secondary Outcome: Percentage of Participants With a Tumor Response
Description: Tumor response was defined as either a complete response or a partial response prior to failure (disease progression, death from any cause, or a second malignancy). A complete response was defined as the complete disappearance on magnetic response imaging of all enhancing tumor and mass effect on a stable or decreasing dose of dexamethasone (or only receiving adrenal replacement doses) accompanied by a stable or improving neurologic examination that was maintained for at least 12 weeks. A partial response was defined as a greater than or equal to 50% reduction in tumor size by bi-dimensional measurement on a stable or decreasing dose of dexamethasone accompanied by a stable or improving neurologic examination that was maintained for at least 12 weeks.
Time Frame: Baseline to the end of the study (up to 20 weeks)
Population: Intent-to-treat population: All enrolled participants who received at least 1 dose of capecitabine.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Capecitabine + Radiation Therapy
Number analyzed (Participants) | 44
Percentage of participants | 2.3 [0.1 to 12.0]

ADVERSE EVENTS:
Time Frame: Adverse events were reported from Baseline up to 30 days after the last treatment (up to 24 weeks).
Description: Safety population: All enrolled participants who received at least 1 dose of capecitabine. One of the 45 participants did not receive treatment and was not included in the safety population.
Arm/Group | Capecitabine + Radiation Therapy
Serious Adverse Events (participants affected / at risk) | 23/44
Other Adverse Events (participants affected / at risk) | 44/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Capecitabine + Radiation Therapy (N=44)
Central nervous system necrosis (Nervous system disorders) | 3
Hydrocephalus (Nervous system disorders) | 3
Convulsion (Nervous system disorders) | 2
Neurological symptom (Nervous system disorders) | 2
Depressed level of consciousness (Nervous system disorders) | 1
Dysarthria (Nervous system disorders) | 1
Haemorrhage intracranial (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Disease progression (General disorders) | 2
Pyrexia (General disorders) | 2
Death (General disorders) | 1
Device malfunction (General disorders) | 1
Irritability (General disorders) | 1
Oedema peripheral (General disorders) | 1
Neutrophil count decreased (Investigations) | 5
White blood cell count decreased (Investigations) | 2
Alanine aminotransferase increased (Investigations) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Dysphagia (Gastrointestinal disorders) | 2
Enterocolitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hypovolaemia (Metabolism and nutrition disorders) | 1
Clostridial infection (Infections and infestations) | 1
Enterocolitis infectious (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Nail infection (Infections and infestations) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Capecitabine + Radiation Therapy (N=44)
Alanine aminotransferase increased (Investigations) | 33
Lymphocyte count decreased (Investigations) | 32
White blood cell count decreased (Investigations) | 27
Platelet count decreased (Investigations) | 25
Blood bilirubin increased (Investigations) | 14
Neutrophil count decreased (Investigations) | 14
Aspartate aminotransferase increased (Investigations) | 11
Weight increased (Investigations) | 11
Gamma-glutamyltransferase increased (Investigations) | 5
Haemoglobin (Investigations) | 4
Weight decreased (Investigations) | 4
Haemoglobin increased (Investigations) | 3
Neutrophil count (Investigations) | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 21
Hypokalaemia (Metabolism and nutrition disorders) | 18
Hypocalcaemia (Metabolism and nutrition disorders) | 17
Hypermagnesaemia (Metabolism and nutrition disorders) | 16
Hyponatraemia (Metabolism and nutrition disorders) | 16
Hyperglycaemia (Metabolism and nutrition disorders) | 15
Hypophosphataemia (Metabolism and nutrition disorders) | 14
Decreased appetite (Metabolism and nutrition disorders) | 11
Hypercalcaemia (Metabolism and nutrition disorders) | 8
Hypernatraemia (Metabolism and nutrition disorders) | 5
Hypoglycaemia (Metabolism and nutrition disorders) | 4
Vomiting (Gastrointestinal disorders) | 35
Nausea (Gastrointestinal disorders) | 15
Constipation (Gastrointestinal disorders) | 14
Abdominal pain (Gastrointestinal disorders) | 11
Diarrhoea (Gastrointestinal disorders) | 11
Stomatitis (Gastrointestinal disorders) | 5
Abdominal distension (Gastrointestinal disorders) | 3
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 16
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 7
Dry skin (Skin and subcutaneous tissue disorders) | 7
Skin exfoliation (Skin and subcutaneous tissue disorders) | 7
Alopecia (Skin and subcutaneous tissue disorders) | 6
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 6
Pruritus (Skin and subcutaneous tissue disorders) | 5
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3
Headache (Nervous system disorders) | 20
Ataxia (Nervous system disorders) | 9
Facial nerve disorder (Nervous system disorders) | 9
VIth nerve disorder (Nervous system disorders) | 8
Hemiparesis (Nervous system disorders) | 6
Dysarthria (Nervous system disorders) | 5
Somnolence (Nervous system disorders) | 4
Vagus nerve disorder (Nervous system disorders) | 4
Central nervous system necrosis (Nervous system disorders) | 3
Dizziness (Nervous system disorders) | 3
Tremor (Nervous system disorders) | 3
Anaemia (Blood and lymphatic system disorders) | 16
Lymphopenia (Blood and lymphatic system disorders) | 9
Leukopenia (Blood and lymphatic system disorders) | 8
Fatigue (General disorders) | 18
Pyrexia (General disorders) | 6
Irritability (General disorders) | 4
Pain (General disorders) | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6
Back pain (Musculoskeletal and connective tissue disorders) | 3
Cushingoid (Endocrine disorders) | 14
Adrenal insufficiency (Endocrine disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3
Anxiety (Psychiatric disorders) | 6
Insomnia (Psychiatric disorders) | 4
Mucosal infection (Infections and infestations) | 8
Pollakiuria (Renal and urinary disorders) | 4
Sinus tachycardia (Cardiac disorders) | 3
Extraocular muscle paresis (Eye disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.